CLINICAL TRIAL: NCT06039124
Title: Subsequent Bevacizumab Treatment in Patients With HHT After the End of BABH Interventional Study. A Descriptive Study.
Brief Title: Subsequent Bevacizumab Treatment in Patients With HHT. Follow up BABH
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1438
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hemorrhagic Hereditary Telangiectasia; HHT
Keywords: HHT; VEGF therapy; BEVACIZUMAB
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HHT patients previously included in BABH study: Clinical and therapeutic follow-up of HHT patients for one year after the end of a clinical trial using bevacizumab.
  Interventions: Other: bevacizumab treatment

INTERVENTIONS:
Other: bevacizumab treatment — Descriptive study of HHT patients (bevacizumab treatment, number of RBC transfused)

SUMMARY:
Bevacizumab is widely prescribed for the treatment of severe bleeding related to epistaxis or gastrointestinal bleeding in HHT.

We studied the efficacy of bevacizumab on severe bleeding in HHT patients in a randomized study recently published (NCT03227263, J Int Med 2023). In this study, 24 patients were included, 12 patients received bevacizumab and 12 patients received placebo. The duration of patient participation was 6 months, including the 2.5-month treatment period and 3.5 month follow-up after treatment.

We describe the evolution of the number of RBC transfused in HHT patients who received bevacizumab during the year after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in BABH study

Exclusion Criteria:

* Patients opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the BABH study (adults, with a confirmed diagnosis of Rendu-Osler disease, presenting with bleeding requiring regular transfusions).
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Bevacizumab treatment description after end of BABH study | 12 months
  Number of patients who received bevacizumab after BABH study. Among patients who received bevacizumab in BABH study: description of re-treatments.
  In patients who received placebo in BABH study: description of treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Service de Médecine Interne et Maladies Vasculaires + Service Neuropédiatrie et neurochirurgie de l'enfant - CHU Angers, Angers
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Montpellier-Hôpital St Eloi, Montpellier

REFERENCES:
- [Derived] Dupuis-Girod S, Decullier E, Riviere S, Lavigne C, Grobost V, Leguy-Seguin V, Maillard H, Chinet T, Fargeton AE, Guilhem A, Hermann R. BEST study: one-year descriptive follow-up of bevacizumab treatment in hereditary haemorrhagic telangiectasia post-BABH interventional study. Ther Adv Hematol. 2025 Apr 14;16:20406207241300828. doi: 10.1177/20406207241300828. eCollection 2025. PMID 40290758